CLINICAL TRIAL: NCT01400594
Title: A Randomized, Double-Blind, Parallel-Group, Multicenter, Placebo-Controlled Study of the Safety & Efficacy of HTU-520 in the Treatment of Mild to Moderate Distal Subungual Onychomycosis of the Toenail
Brief Title: Safety & Efficacy Study of HTU-520 in the Treatment of Distal Subungual Onychomycosis of the Toenail
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hisamitsu Pharmaceutical Co., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HTU-520-US01
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-05

CONDITIONS: Onychomycosis
Keywords: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HTU-520 Patch (Experimental): Subjects will receive HTU-520 patch in a 1:1 ratio for 48 weeks applied to all toenails.
  Interventions: Drug: HTU-520 Patch
- Placebo Patch (Placebo Comparator): Subjects will receive placebo patch in a 1:1 ratio for 48 weeks applied to all toenails.
  Interventions: Other: Placebo Patch

INTERVENTIONS:
Drug: HTU-520 Patch — Terbinafine hydrochloride patch
  Other Names: HTU-520
  Arms: HTU-520 Patch
Other: Placebo Patch — Treatment with Placebo Patch
  Other Names: Sham treatment
  Arms: Placebo Patch

SUMMARY:
This is a multicenter, randomized, double-blind, parallel-group, placebo-controlled study of HTU-520 in subjects with clinically diagnosed onychomycosis of the great toenail.

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Parallel-Group, Multicenter, Placebo-Controlled Study of the Safety & Efficacy of HTU-520 in the Treatment of Mild to Moderate Distal Subungual Onychomycosis of the Toenail

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of DSO for at least one great toenail
2. Direct microscopy of subungual debris positive for hyphal elements (KOH test)
3. Culture confirmation of the growth of a dermatophyte
4. Good general health
5. Willing to refrain from using any lotions, creams, liquids, or polish on treated toenails
6. Willing to refrain from receiving pedicures for the duration of the study
7. If female, using an acceptable form of birth control

Exclusion Criteria:

1. Unable to apply test product onto toenails by him/herself
2. Use of topical antifungal agents on the nail within 1 month
3. Uncontrolled diabetes
4. Onychomycosis of the fingernails
5. Confirmed non-dermatophyte infection of the target toenail
6. Structural deformities of the target toenail, open wounds, lesions, sores, surgery on the feet or toenails
7. History of severe or chronic immunosuppression, an immunocompromised condition
8. Any systemic or dermatologic disorder, such as severe eczema, or severe atopic dermatitis
9. Psoriasis of the toenails
10. Hypersensitivity or allergy to topical preparations (including terbinafine) or adhesive dressings

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2011-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Determination of status with respect to complete cure (mycological cure together with clinical cure) of onychomycosis of the toenail. | 48 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Donald Sislen, MD, Principal Investigator; Susan Taylor, MD, Principal Investigator; Melanic Appell, MD, Principal Investigator; Harry I. Geisberg, MD, Principal Investigator; Michele D. Reynolds, MD, Principal Investigator; Linda P. Murray, MD, Principal Investigator; Michael P. Kyle, MD, Principal Investigator; Kenneth W. Dawes, MD, Principal Investigator; Hassan Malik, MD, Principal Investigator; Francisco A. Kerdel, MD, Principal Investigator; Leon Kircik, MD, Principal Investigator; Mark S. Nestor, MD, Principal Investigator; Douglas N. Robins, MD, Principal Investigator; Pranav B. Sheth, MD, Principal Investigator; Martin Throne, MD, Principal Investigator; Patrick S. Agnew, MD, Principal Investigator; David Bolshoun, MD, Principal Investigator; Gordon T. Connor, MD, Principal Investigator; Boni Elewski, MD, Principal Investigator; Laura Ferris, MD, Principal Investigator; Steven E. Kempers, MD, Principal Investigator; Daniel G. Lorch, MD, Principal Investigator; James A. Solomon, MD, Principal Investigator; Norman Bystol, MD, Principal Investigator; William P. Coleman, MD, Principal Investigator; Paul Gillum, MD, Principal Investigator; William P. Jennings, MD, Principal Investigator; Ramin Farsad, MD, Principal Investigator; Jeffrey C. Noroyan, MD, Principal Investigator; Fredric S. Brandt, MD, Principal Investigator; Robert Dunne, MD, Principal Investigator; Marta Rendon, MD, Principal Investigator; Kimball W Silverton, DO, Principal Investigator; John Tassone, DPM, Principal Investigator
Locations (37):
- United States (37):
  - Total Skin and Beauty Dermatology Center, Birmingham, Alabama
  - Radiant Research, Inc., Birmingham, Alabama
  - UAB Department of Dermatology, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Clinical Research Advantage, Inc., Glendale, Arizona
  - Radiant Research, Inc., Tucson, Arizona
  - Diagnamics, Inc., Encinatas, California
  - Radiant Research, Inc., Denver, Colorado
  - Center for Clinical and Cosmetic Research, Aventura, Florida
  - Marta Rendon, MD, Skin Care Research, Inc., Boca Raton, Florida
  - Pab Clinical Research, Brandon, Florida
  - Dermatology Research Institute, Coral Gables, Florida
  - Ameriderm Research, Jacksonville, Florida
  - Lake Washington Foot & Ankle Center, Melbourne, Florida
  - Florida Academic Dermatology Center, Miami, Florida
  - Ameriderm Research, Ormond Beach, Florida
  - Leavitt Medical Associates ofFL, Ormond Beach, Florida
  - Radiant Research, Inc., Pinellas Park, Florida
  - Radiant Research, Inc., Atlanta, Georgia
  - Radiant Research, Inc., Chicago, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Derm Research, LLC, Louisville, Kentucky
  - William P Coleman III, MD, Metairie, Louisiana
  - Callender center for Clinical Research, Glenn Dale, Maryland
  - Assoc Foot Clinic & Surgery Specialists, Flint, Michigan
  - Silverton Skin Institute, Grand Blanc, Michigan
  - University of Minnesota, Minnesota Clinical Study Center, Fridley, Minnesota
  - Radiant Research, St Louis, Missouri
  - Radiant Research, Inc., Akron, Ohio
  - Group Health Associates, Tri-Health, Cincinnati, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Society Hill Dermatology, Philadelphia, Pennsylvania
  - University of Pittsburg Medical Center, Department of Dermatology, Pittsburgh, Pennsylvania
  - Radiant Research, Inc., Anderson, South Carolina
  - Radiant Research, Inc., Dallas, Texas
  - Radiant Research, Inc., San Antonio, Texas
  - Coastal Podiatry Group, Virginia Beach, Virginia